CLINICAL TRIAL: NCT03217409
Title: A Multicenter Clinical Trial to Compare the Efficacy and Safety Between Rosuvastatin/Ezetimibe Combination and Monotherapy of Rosuvastatin in Patients With Diabetes Mellitus and Hypercholesterolemia
Brief Title: A Study to Compare Rosuvastatin/Ezetimibe and Rosuvastatin in Patients With Diabetes Mellitus and Hypercholesterolemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Collaborators: Linical Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC022
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus and Hypercholesterolemia
MeSH Terms: conditions — Diabetes Mellitus; Hypercholesterolemia | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvastatin+Ezetimibe (Experimental): Rosuvastatin 5mg+Ezetimibe 10mg Rosuvamibe ® Tablet, 1T, Once a day/8week
  Interventions: Drug: Rosuvastatin+Ezetimibe
- Rosuvastatin (Active Comparator): Rosuvastatin 5mg Monorova ® Tablet, 1T, Once a day/8week
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin+Ezetimibe — Rosuvastatin 5mg+Ezetimibe 10mg
  Other Names: Rosuvamibe ® 10/5mg
  Arms: Rosuvastatin+Ezetimibe
Drug: Rosuvastatin — Rosuvastatin 5Mg Tablet
  Other Names: Monorova ® 5mg
  Arms: Rosuvastatin

SUMMARY:
A Study to Compare Rosuvastatin/Ezetimibe Combination and Monotherapy in Patients with Diabetes Mellitus and Hypercholesterolemia.

DETAILED DESCRIPTION:
This trial is conducted to compare the efficacy and safety between Rosuvastatin/Ezetimibe combination and Rosuvastatin monotherapy in patients with Diabetes Mellitus and Hypercholesterolemia for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 19 or ≤ 75 years of age
* Subjects undergoing treatment for type 2 diabetes
* Subjects undergoing treatment of statin for hypercholesterolemia
* Fasting LDL-C ≤ 250mg/dL at the screening visit
* Fasting LDL-C ≥70mg/dL or ≤ 160mg/dL at the randomization visit
* Fasting TG<500mg/dL

Exclusion Criteria:

* Subjects with hypersensitivity reaction to Statin and Ezetimibe
* Subjects with severe kidney disease
* Subjects with HIV positive result at the screening
* Pregnant or breast-feeding subjects
* Subjects with taking any medication affecting level of LDL (Fenofibrate, Omega 3 fatty aicd etc.)
* Insulin-treated Subjects
* Other exclusions applied

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Low density lipoprotein cholesterol (LDL-C) (%) | baseline, Week 8
  The rate of change(%) of LDL-C at Week 8 compared to the baseline

SECONDARY OUTCOMES:
Low density lipoprotein cholesterol (LDL-C) (100mg/dL) | baseline, Week 8
  The ratio of patients who reached the treatment target (100mg/dL) of LDL-C at Week 8 compared to the baseline
HbA1C, Glycated albumin, Homeostasis model assessment Insulin resistance(HOMA-IR), Homeostasis model assessment ß cell(HOMA-ß) resistance(HOMA-IR), Homeostasis model assessment ß cell(HOMA-ß) | baseline, Week 8
  Variation of HbA1C, Glycated albumin, Homeostasis model assessment Insulin resistance(HOMA-IR), Homeostasis model assessment ß cell(HOMA-ß) at Week 8 compared to the baseline resistance(HOMA-IR), Homeostasis model assessment ß cell(HOMA-ß) change form the baseline at Week 8
LDL-C, Non HDL-C, HDL-C, Triglyceride(TG), Total cholesterol(TC), Apolipoprotein A1, Apolipoprotein B, Lipid ratios (LDL-C/HDL-C, TC/HDL-C, Non- HDL-C/HDL-C) Apolipoprotein A1, Apolipoprotein B, Lipid ratios (LDL-C/HDL-C, TC/HDL-C, Non- HDL-C/HDL-C) | baseline, Week 8
  Variation of LDL-C, Non HDL-C, HDL-C, Triglyceride(TG), Total cholesterol(TC), Apolipoprotein A1, Apolipoprotein B, Lipid ratios (LDL-C/HDL-C, TC/HDL-C, Non- HDL-C/HDL-C) at Week 8 compared to the baseline Apolipoprotein A1, Apolipoprotein B, Lipid ratios (LDL-C/HDL-C, TC/HDL-C, Non- HDL-C/HDL-C) change form the base line at Week 8
Thiobarbituric acid reactive substances(TBARs) | baseline, Week 8
  Absolute value change of Thiobarbituric acid reactive substances(TBARs) at Week 8 compared to baseline to baseline.
Fibroblast Growth Factor 21 | baseline, Week 8
  Absolute value change of Fibroblast Growth Factor 21 at Week 8 compared to baseline.

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Soon Chun Hyang University Hospital Gumi, Gumi
  - Soon Chun Hyang University Hospital Bucheon, Gyeonggi-do
  - Soon Chun Hyang University Hospital Seoul, Seoul

IPD SHARING:
Plan to Share IPD: No